CLINICAL TRIAL: NCT02638740
Title: To Assess the Efficacy of Mustard Oil and Salt Massage as an Adjunct to Scaling and Root Planing in Patients With Chronic Periodontitis: A Clinical Study
Brief Title: To Study the Beneficial Effect of Mustard Oil and Salt Massaging With Oral Prophylaxis in Patients With Gum Diseases
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Government College of Dentistry, Indore (Other)
Responsible Party: Principal Investigator, Dr. Trishna Mhapsekar, Dr., Government College of Dentistry, Indore
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GDCIndore
Record Dates: First submitted 2015-12-20; First posted 2015-12-23 (Estimated); Last update posted 2017-04-18 (Actual); Status verified 2017-04

CONDITIONS: Chronic Periodontitis
MeSH Terms: conditions — Chronic Periodontitis | interventions — Tooth Exfoliation; Root Planing; mustard oil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- SCALING AND ROOT PLANING (SRP) (Active Comparator): Scaling and root planning with ultrasonic scalar
  Interventions: Procedure: SCALING AND ROOT PLANING (SRP)
- MUSTARD OIL AND SALT MASSAGE WITH SRP (Experimental): Scaling and root planing was done with ultrasonic scalar. It was followed by gum massaging with 0.32gm salt in 5ml mustard oil for 5min, twice daily for 90 days.
  Interventions: Procedure: SCALING AND ROOT PLANING (SRP); Procedure: MUSTARD OIL AND SALT MASSAGE WITH SRP

INTERVENTIONS:
Procedure: SCALING AND ROOT PLANING (SRP) — Scaling and root planning done with ultrasonic scalar with reinforcement of oral hygiene measures and follow up for 90 days.
Procedure: MUSTARD OIL AND SALT MASSAGE WITH SRP — Scaling and root planing was done with ultrasonic scalar. It was followed by gum massaging with 0.32gm salt in 5ml mustard oil for 5min, twice daily for 90 days.
  Arms: MUSTARD OIL AND SALT MASSAGE WITH SRP

SUMMARY:
Periodontal disease is a chronic inflammatory process accompanied by destruction of Periodontium, and sometimes loss of teeth. Periodontal disease is highly prevalent especially in developing and underdeveloped countries affecting more than 80% population. Epidemiological studies have shown that about 10% of the adult population suffer from severe periodontitis (Brown et al. 1990, Gjermo 1998). Studies indicate that the periodontal lesion is not strictly a localized process but may lead to systemic alterations in immune system. Various studies confirm the microbial etiology of periodontal disease.

DETAILED DESCRIPTION:
Periodontal disease is a chronic inflammatory process accompanied by destruction of Periodontium, and sometimes loss of teeth. Periodontal disease is highly prevalent especially in developing and underdeveloped countries affecting more than 80% population. Epidemiological studies have shown that about 10% of the adult population suffer from severe periodontitis (Brown et al. 1990, Gjermo 1998). Studies indicate that the periodontal lesion is not strictly a localized process but may lead to systemic alterations in immune system. Various studies confirm the microbial etiology of periodontal disease. The bacteria that cause periodontitis include mainly diversity of anerobic bacteria; Porphyromonas Gingivalis, Fusobacterium Nucleatum, Peptostreptococcus, Prevotella species being the most significant.

Various therapeutic approaches are available for treatment of this disease utilizing non surgical and surgical methods, but the treatment is still challenging for the clinician and cumbersome for the patients. In many cases of moderate to severe chronic periodontitis anti- inflammatory and antibiotics are used as an adjunct. Systemic antibiotic agents may reduce or eliminate microbes that cannot be removed by Scaling and Root Planing. This includes microbes that have penetrated tissues or root surfaces which may act as reservoir for recolonization. However synthetic antibiotics and anti-inflammatory agents result in complications like drug resistance, gastrointestinal complications, congestive heart failures and renal failures and other complications.

Especially in India Mustard Oil and Salt is long being used for gum massage and for maintenance and improvement of Oral Hygiene. As this practice of using homemade formulation is beneficial for Gingival and Periodontal health, economic and free from any major side effects it should be studied to document its efficacy as an adjunct to Scaling and Root Planing. Mustard oil is considered to have low saturated fat. The monounsaturated fatty acids and proper ratio of polyunsaturated fatty acids improve heart health, lowers triglyceride, prevents obesity. Massage with mustard oil relieves rheumatism and arthritis, sprains and aches. The selenium present in the oil reduces effects of asthma and joint pain. High level of Vit. E improves skin health and impart protection against UV rays. Mustard seeds are effective in gastrointestinal and colorectal cancer, as mustard is rich in glucosinolate and phytonutrients. It is effective in curing cold, cough, body pains & aches. Salt in topical formulation is found to have anti inflammatory action.Hence this study aims to evaluate this versatile formulation in treatment of Chronic Periodontitis. As the use of Mustard Oil and Salt is practiced by a strata of population in our country thus it is advisable and necessary to assess scientifically the efficacy of mustard oil and salt massage in improving Gingival and Periodontal Health.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with moderate to severe Chronic Generalized Periodontitis
* Not undergone any major periodontal treatment in past 6 months
* Otherwise clinically healthy patients

Exclusion Criteria:

* Any known systemic diseases specially Diabetes and other major diseases.
* Patients on anti-inflammatory drugs or antibiotics
* Patient allergic to any material used for the study
* Pregnant and lactating mothers
* Periodontal therapy in past 6 months
* Smoker and tobacco chewer

Ages: 28 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2015-06; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Plaque Index (Turesky modification of Quigely Hein Index, 1970) | Baseline
  2 surfaces of all tooth measured

SECONDARY OUTCOMES:
Plaque Index (Turesky modification of Quigely Hein Index, 1970) | 1 week
  2 surface of each tooth measured
Plaque Index (Turesky modification of Quigely Hein Index, 1970) | 2 week
  2 surface of each tooth measured
Plaque Index (Turesky modification of Quigely Hein Index, 1970) | 4 week
  2 surface of each tooth measured
Plaque Index (Turesky modification of Quigely Hein Index, 1970) | 8 week
  2 surface of each tooth measured
Plaque Index (Turesky modification of Quigely Hein Index, 1970) | 12 week
  2 surface of each tooth measured
Probing pocket depth (PPD) | Baseline
  6 surface of each tooth measured
Probing pocket depth (PPD) | 1 week
  6 surface of each tooth measured
Probing pocket depth (PPD) | 2 week
  6 surface of each tooth measured
Probing pocket depth (PPD) | 4 week
  6 surface of each tooth measured
Probing pocket depth (PPD) | 8 week
  6 surface of each tooth measured
Probing pocket depth (PPD) | 12 week
  6 surface of each tooth measured
Modified Gingival Index (Lobene, Weather, Ford, Ross, Lamm, 1986) | Baseline
  4 sites of all tooth measured
Modified Gingival Index (Lobene, Weather, Ford, Ross, Lamm, 1986) | 1 week
  4 sites of all tooth measured
Modified Gingival Index (Lobene, Weather, Ford, Ross, Lamm, 1986) | 2 week
  4 sites of all tooth measured
Modified Gingival Index (Lobene, Weather, Ford, Ross, Lamm, 1986) | 4 week
  4 sites of all tooth measured
Modified Gingival Index (Lobene, Weather, Ford, Ross, Lamm, 1986) | 8 week
  4 sites of all tooth measured
Modified Gingival Index (Lobene, Weather, Ford, Ross, Lamm, 1986) | 12 week
  4 sites of all tooth measured
Clinical Attachment Level (CAL) | Baseline
  6 surfaces of each teeth measured
Clinical Attachment Level (CAL) | 1 week
  6 surfaces of each teeth measured
Clinical Attachment Level (CAL) | 2 week
  6 surfaces of each teeth measured
Clinical Attachment Level (CAL) | 4 week
  6 surfaces of each teeth measured
Clinical Attachment Level (CAL) | 8 week
  6 surfaces of each teeth measured
Clinical Attachment Level (CAL) | 12 week
  6 surfaces of each teeth measured
Mobility Index (S.C Miller 1974) | Baseline
  Mobility of each tooth measured
Papillary Bleeding Index (Saxer and Muhlemann, 1975) | Baseline
  Interdental papilla of each teeth in checked
Papillary Bleeding Index (Saxer and Muhlemann, 1975) | 1 week
  Interdental papilla of each teeth in checked
Papillary Bleeding Index (Saxer and Muhlemann, 1975) | 2 week
  Interdental papilla of each teeth in checked
Papillary Bleeding Index (Saxer and Muhlemann, 1975) | 4 week
  Interdental papilla of each teeth in checked
Papillary Bleeding Index (Saxer and Muhlemann, 1975) | 8 week
  Interdental papilla of each teeth in checked
Papillary Bleeding Index (Saxer and Muhlemann, 1975) | 12 week
  Interdental papilla of each teeth in checked
Russels Periodontal Index | Baseline
  Each tooth measure

CONTACTS AND LOCATIONS:
Overall Officials: trishna Mhapsekar, Principal Investigator — Government College of Dentistry, Indore
Locations (1):
- Govt. College of Dentistry Indore, M.P. India, Indore, M.P, India

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Quist SR, Wiswedel I, Quist J, Gollnick HP. Anti-inflammatory effects of topical formulations containing sea silt and sea salt on human skin in vivo during cutaneous microdialysis. Acta Derm Venereol. 2011 Sep;91(5):597-9. doi: 10.2340/00015555-1128. No abstract available. PMID 21597673
- [Background] Singla N, Acharya S, Martena S, Singla R. Effect of oil gum massage therapy on common pathogenic oral microorganisms - A randomized controlled trial. J Indian Soc Periodontol. 2014 Jul;18(4):441-6. doi: 10.4103/0972-124X.138681. PMID 25210256
- [Background] Fourel J, Falabregues R, Bonfil JJ. A clinical approach to gingival stimulation. J Periodontol. 1981 Mar;52(3):130-4. doi: 10.1902/jop.1981.52.3.130. PMID 6939833